CLINICAL TRIAL: NCT04032353
Title: Medical Consortium for Screening Upper Gastrointestinal Cancers With Magnetically Controlled Capsule Gastroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yanqing Li (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, vice president of Qilu Hospital, Shandong University
Organization: Shandong University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019SDU-QILU-150
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Capsule Endoscopy; Cancer of Stomach; Cancer of Esophagus; Health Policy
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical Consortium (Other): subjects involved in medical consortium for screening upper gastrointestinal canccers(MCSC)
  Interventions: Other: Medical Consortium

INTERVENTIONS:
Other: Medical Consortium — subjects received intensive follow-up by coordinators according to the predifined protocol of MCSC

SUMMARY:
The aim of our study was to demonstrate the efficacy and feasibility of the medical consortium for screening upper gastrointestinal cancers with magnetically controlled capsule gastroscopy.

DETAILED DESCRIPTION:
In this study, the investigators designed a propective cohort study to evaluate the the efficacy and feasibility of medical consortium for screening upper gastrointestinal cancers (MCSC) with magnetically controlled capsule gastroscopy (MCCG).

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic subjects undergong magnetically controlled capsule gastroscopy for health checkup in medical consotium;
* subjects able to give informed consent

Exclusion Criteria:

* suspected or known intestinal stenosis, obstruction, or fistula;
* inoperability of refusal to accept any abdominal surgery;
* dysphagia or gastric paralysis;
* previous history of gastrointestinal disease;
* with pacemaker, implanted-cardiac defibrillator or other implanted electromedical devices;
* need for standard magnetic resonance imaging examination within seven days after swallowing the MCCG, unless the capsule is confirmed to have been excreted;
* other factors that are not suitable for inclusion evaluated by medical stuff

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10000 (Estimated)
Dates: Start 2018-12-31 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of upper gastrointestinal cancers, including gastric cancer and esophageal cancer. | 12 months

SECONDARY OUTCOMES:
tthe focal lesions of upper gastrointestinal tract | 12 months

OTHER OUTCOMES:
adverse events | 12 months
  safety assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China